CLINICAL TRIAL: NCT02057484
Title: A Long-term Follow-up of Adult Kidney and Liver Allograft Recipients Previously Enrolled Into a Tacrolimus (Advagraf) Trial. A Multicentre Non-interventional Post Authorization Study (PAS)
Brief Title: A 5 Year Follow-up of Patients Who Were Previously Enrolled Into an Advagraf Trial Following a Liver or Kidney Transplant
Acronym: ADDRESS
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: PMR-EC-1213
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplant; Kidney Transplant
Keywords: long-term follow-up; liver transplant; kidney transplant; Advagraf; Tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Organ transplant patients treated with Advagraf: To evaluate long-term graft survival in patients treated with Advagraf
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Advagraf

SUMMARY:
The purpose of this study is to evaluate the impact of Advagraf, prolonged-release, once daily tacrolimus formulation, on long-term graft survival in kidney and liver allograft recipients. This study will also evaluate the overall long-term impact of Advagraf on kidney and liver allograft recipients.

DETAILED DESCRIPTION:
Prograf is one of the medications taken by a patient after they have had a liver or kidney transplant to prevent their body from rejecting the new liver or kidney transplant. Prograf is taken by the patient twice a day. Advagraf is a similar medication but is taken by the patient only once a day. There is some evidence emerging that may show that this once-a-day medication may show additional benefits over the twice a day medication, such as, patients more likely to remember to take this medication. Also, this once a day medication is slowly released in the body through the course of a day which in turn may provide better protection against the body rejecting the new transplanted organ over a longer period.

This study will follow up adult patients who were previously enrolled in an Advagraf trial after they have had a liver or kidney transplant. The information collected for this study will be information that the patient's doctor will normally collect when he/she sees the patient for their regular check-ups. Information will be collected once a year for a period of 5 years from when the patient received their new organ transplant. It is hoped that patient information collected during the study will provide prescribers with useful information in treatment of organ transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Participated in one of the selected Astellas sponsored clinical trials :

  * DIAMOND - PMR-EC-1106
  * ADVANCE - PMR-EC-1211
  * ADHERE - PMR-EC-1212
  * Or, any potential new Astellas-sponsored Advagraf trial
* Assigned to treatment with Advagraf in one of the selected Astellas sponsored clinical trials and received a kidney or liver organ transplant.

NOTE: The primary objective is to study long-term graft survival in patients currently or previously treated with Advagraf. Therefore patients do not have to be currently receiving Advagraf to be included, nor do they have to have completed a previous Astellas clinical trial.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had previously participated in the following Astellas sponsored clinical trial also known as "feeder trials":
  DIAMOND / PMR-EC1106 ADVANCE / PMR-EC-1211 ADHERE / PMR-EC-1212 Any potential new Astellas-sponsored Advagraf trial
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Overall graft survival (time to graft loss) | Annually from date of transplant and for 5 five years
  At each annual visit there will be a simple assessment to determine if the graft has survived or not.

SECONDARY OUTCOMES:
Overall patient survival | Annually from date of transplant and for 5 five years
  At each annual visit there will be a simple assessment to determine if the patient has survived or not.
Renal Function | Annually from date of transplant and for 5 five years
  At each annual visit serum creatinine results, which is part of routine clinical practice will be collected from the patient's medical records. This will be used by the sponsor to calculate estimated glomerular filtration rate.
Emergence of de novo Donor Specific Antibody | Annually from date of transplant and for 5 five years
  If the site collects this information as part of routine clinical practice, only then will this information be collected.
Biopsy proven acute rejection episodes | Annually from date of transplant and for 5 five years
  All rejection episodes captured in the medical records of the patient from one annual visit to the next will be collected for this study
Immunosuppression regimen | Annually from date of transplant and for 5 five years
  Any immunosuppression regimen, doses and changes in doses from one annual visit to another, as well any annual trough levels of tacrolimus.
Medical conditions of interest | Annually from date of transplant and for 5 five years
  Medical conditions of interest include, diabetes mellitus, and cardiovascular conditions such as myocardial infarction and strokes.
Infections of interest | Annually from date of transplant and for 5 five years
  Infections of interest include cytomegalovirus and BK virus

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe Ltd.
Locations (145):
- Austria (3):
  - Site AT43001, Innsbruck
  - Site AT43003, Linz
  - Site AT43002, Vienna
- Site BY37501, Minsk, Belarus
- Belgium (7):
  - Site BE32007, Brussels, Brussels Capital
  - Site BE32002, Brussels
  - Site BE32001, Ghent
  - Site BE32003, Leuven
  - Site BE32005, Leuven
  - Site BE32008, Liège
  - Site BE32009, Liège
- Canada (2):
  - Site CA15001, Halifax, Nova Scotia
  - Site CA15003, Montreal, Quebec
- Czechia (6):
  - Site CZ42006, Brno
  - Site CZ42004, Hradec Králové
  - Site CZ42003, Olomouc
  - Site CZ42005, Ostrava
  - Site CZ42001, Prague
  - Site CZ42002, Prague
- Site EE37201, Tartu, Estonia
- Finland (2):
  - Site FI35801, Helsinki
  - Site FI35802, Helsinki
- France (28):
  - Site FR33020, Angers
  - Site FR33007, Besançon
  - Site FR33012, Bordeaux
  - Site FR33025, Brest
  - Site FR33027, Clermont-Ferrand
  - Site FR33003, Clichy, Paris
  - Site FR33001, Créteil
  - Site FR33029, Créteil
  - Site FR33032, Dijon
  - Site FR33026, Le Kremlin-Bicêtre
  - Site FR33018, Limoges
  - Site FR33011, Marseille
  - Site FR33014, Montpellier
  - Site FR33023, Nantes
  - Site FR33004, Nice
  - Site FR33015, Nice
  - Site FR33008, Paris
  - Site FR33010, Paris
  - Site FR33031, Paris
  - Site FR33019, Paris
  - Site FR33024, Rouen
  - Site FR33022, Saint-Etienne
  - Site FR33017, Strasbourg
  - Site FR33034, Toulouse
  - Site FR33009, Tours
  - Site FR33030, Tours
  - Site FR33028, Vandœuvre-lès-Nancy
  - Site FR33002, Villejuif
- Germany (19):
  - Site DE49011, Aachen
  - Site DE49004, Berlin
  - Site DE49019, Bochum
  - Site DE49013, Düsseldorf
  - Site DE49030, Essen
  - Site DE49001, Frankfurt am Main
  - Site DE49014, Halle
  - Site DE49022, Hannoversch Münden
  - Site DE49005, Hanover
  - Site DE49018, Hanover
  - Site DE49008, Jena
  - Site DE49015, Kaiserslautern
  - Site DE49002, Kiel
  - Site DE49027, Mannheim
  - Site DE49025, Munich
  - Site DE49016, Munich
  - Site DE49010, Regensburg
  - Site DE49017, Rostock
  - Site DE49006, Tübingen
- Hungary (3):
  - Site HU36001, Budapest
  - Site HU36003, Debrecen
  - Site HU36002, Szeged
- Site IE35301, Dublin, Ireland
- Italy (19):
  - Site IT39015, Ancona
  - Site IT39003, Bergamo
  - Site IT39005, Bologna
  - Site IT39013, Bologna
  - Site IT39006, Genova
  - Site IT39014, L’Aquila
  - Site IT39012, Milan
  - Site IT39009, Milan
  - Site IT39008, Naples
  - Site IT39002, Padua
  - Site IT39010, Padua
  - Site IT39016, Palermo
  - Site IT39004, Rome
  - Site IT39020, Rome
  - Site IT39017, Salerno
  - Site IT39019, Siena
  - Site IT39021, Treviso
  - Site IT39001, Udine
  - Site IT39011, Vicenza
- Site LV37101, Riga, Latvia
- Site NL31001, Maastricht, Netherlands
- Poland (6):
  - Site PL48003, Gdansk
  - Site PL48006, Katowice
  - Site PL48005, Lodz
  - Site PL48007, Poznan
  - Site PL48004, Szczecin
  - Site PL48001, Warsaw
- Site PT35102, Lisbon, Portugal
- Romania (2):
  - Site RO40001, Bucharest
  - Site RO40003, Bucharest
- Russia (9):
  - Site RU70014, Kemerovo
  - Site RU70005, Moscow
  - Site RU70002, Moscow
  - Site RU70004, Moscow
  - Site RU70007, Moscow
  - Site RU70010, Omsk
  - Site RU70011, Volzhskiy
  - Site RU70013, Volzhskiy
  - Site RU70012, Yekaterinburg
- Slovakia (2):
  - Site SK42101, Banská Bystrica
  - Site SK42102, Bratislava
- South Korea (5):
  - Site KR82007, Busan
  - Site KR82006, Daegu
  - Site KR82002, Seoul
  - Site KR82005, Seoul
  - Site KR82001, Seoul
- Spain (19):
  - Site ES34001, L'Hospitalet de Llobregat, Barcelona
  - Site ES34019, Barakaldo, Vizcaya
  - Site ES34005, A Coruña
  - Site ES34017, Alicante
  - Site ES34012, Badalona-Barcelona
  - Site ES34004, Barcelona
  - Site ES34011, Barcelona
  - Site ES34003, Barcelona
  - Site ES34010, Córdoba
  - Site ES34018, L'Hospitalet de Llobregat
  - Site ES34006, Madrid
  - Site ES34013, Madrid
  - Site ES34015, Madrid
  - Site ES34009, Santa Cruz de Tenerife
  - Site ES34020, Santander
  - Site ES34014, Seville
  - Site ES34021, Valencia
  - Site ES34016, Valladolid
  - Site ES34007, Zaragoza
- Sweden (3):
  - Site SE46001, Gothenburg
  - Site SE46002, Stockholm
  - Site SE46004, Uppsala
- Site CH41002, Bern, Switzerland
- United Kingdom (3):
  - Site GB44001, Birmingham
  - Site GB44003, Leeds
  - Site GB44002, London

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results Web site — https://astellasclinicalstudyresults.com/study.aspx?ID=278